CLINICAL TRIAL: NCT00279084
Title: Prospective Randomized Controlled Open-Labelled Trial Comparing Effect of Two Haemoglobin Levels (110- 129 g/L and 130 - 149 g/L) on Progression of Chronic Kidney Disease in Patients With Type 2 Diabetes and With Chronic Kidney Disease
Brief Title: NEPHRODIAB2 Prospective Randomized Controlled Open-Labelled Trial Comparing Effect of Two Haemoglobin Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2003.315
Record Dates: First submitted 2006-01-18; First posted 2006-01-19 (Estimated); Last update posted 2007-10-04 (Estimated); Status verified 2007-10

CONDITIONS: Chronic Kidney Disease
Keywords: Anaemia; Chronic kidney disease; Type 2 diabetes; Randomized trial
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia; Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: GROUP A: if necessary, martial treatment and / or erythropoietin treatment to achieve the goal of haemoglobin level from 110 to 129 g/L.
Drug: GROUP B: martial treatment and / or erythropoietin treatment to achieve the goal of haemoglobin level from 130 to 149 g/L

SUMMARY:
In type 2 diabetics, progression from chronic kidney disease to end stage renal disease may be slowed down by therapeutic interventions as angiotensin converting enzyme inhibitors use, control of high blood pressure and proteinuria, control of hyperglycaemia, protein intake restriction, smoking cessation.

Correcting anaemia in these patients may prevent impairment of renal function. International guidelines indicate that haemoglobin level has to be of 110 g/L in these patients. We conduct an interventional randomized trial to evaluate the potential benefit of an haemoglobin level of 130 g/L in patients with type 2 diabetes and with a chronic kidney disease defined by a Cockcroft's creatinine clearance of 25 - 60 ml/min.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes. Age between 18 and 80 years, male or female. Cockcroft's clearance between 25 and 60 ml / min. Haemoglobin level superior to 100 g/L and strictly inferior to 130 g/L

Exclusion Criteria:

Malignancy Solid organ transplant Acute pathology in the two months before inclusion date Myocardial infarction, stroke, pulmonary embolism in the six months before inclusion date Contra-indication to martial treatment or EPO treatment Present inclusion in another clinical study Patient who cannot answer questions of SF36 questionnaire

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204
Dates: Start 2004-01

PRIMARY OUTCOMES:
Decrease in Cockcroft's creatinine clearance between inclusion and end of two years follow-up period.

SECONDARY OUTCOMES:
Death
Angina
Stroke
Peripheral acute ischemia, vascular angioplasty, surgical vascular bypass, amputation
Heart failure
Pulmonary embolism
Deep venous thrombosis and haemodialysis fistula thrombosis
Bacterial infectious disease
Renal replacement therapy (dialysis or pre-emptive renal transplantation)
Quality of life: SF 36 auto-questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel VILLAR, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Joëlle Gillet, Lyon, France

REFERENCES:
- [Derived] Villar E, Lievre M, Kessler M, Lemaitre V, Alamartine E, Rodier M, Francois M, Zaoui P, Moranne O, Choukroun G, Guerraoui A, Jolivot A, Janin G, Branger B, Heng AE, Boudray C, Bissery A, Rabilloud M, Pouteil-Noble C. Anemia normalization in patients with type 2 diabetes and chronic kidney disease: results of the NEPHRODIAB2 randomized trial. J Diabetes Complications. 2011 Jul-Aug;25(4):237-43. doi: 10.1016/j.jdiacomp.2011.03.003. Epub 2011 May 20. PMID 21601481